CLINICAL TRIAL: NCT03130803
Title: Biomarkers of Insufficient Sleep and Sleepiness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Kenneth Wright, Professor, University of Colorado, Boulder
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: R01HL132150 (NIH)
Record Dates: First submitted 2017-04-21; First posted 2017-04-27 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Sleep Deprivation; Insufficient Sleep Syndrome; Sleep Wake Disorders
MeSH Terms: conditions — Sleep Deprivation; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (No Intervention): 9 hour sleep opportunity at habitual sleep/wake times for 14 days at home and 1 day in lab repeated for visit 1 and visit 2
- Insufficient Sleep (Experimental): 2 days with 5 hour sleep opportunities immediately following baseline on both visit 1 and visit 2.
  Interventions: Behavioral: Insufficient Sleep

INTERVENTIONS:
Behavioral: Insufficient Sleep — 2 days with 5 hour sleep opportunity per day
  Arms: Insufficient Sleep

SUMMARY:
Sleep and wakefulness disorders impact 50 to 70 million Americans and insufficient sleep is epidemic with over 50% of Americans reporting less than 7 hours of sleep per night. Health problems associated with insufficient sleep include inflammation, depression and anxiety, diabetes, stress, drug abuse, poor quality of life, obesity, and fatigue related accidents on the job/while driving. While the contribution of sleep to overall health, well-being, and public safety is recognized, no established clinical biomarkers of sleep deficiency exist. Such biomarkers would have utility as road-side biomarkers of sleepiness (e.g., drowsy driving), monitoring on the job fatigue/fitness for duty (e.g., transportation, military ops health care), monitoring sleep health, as well as for clinical diagnostics and measures of clinical treatment outcomes. Thus, investigators designed a controlled laboratory insufficient sleep protocol utilizing metabolomics to identify biomarkers of insufficient sleep. Investigators propose to identify changes in metabolites that consistently occur during insufficient sleep. As an exploratory outcome investigators will examine associated changes in metabolites and cognitive performance during insufficient sleep.

DETAILED DESCRIPTION:
Impaired sleep affects millions of people each year representing an important public health issue. This project will utilize metabolomics approaches to identify biomarkers in the blood that respond consistently to insufficient sleep. The overall goal of this project is to use a discovery and targeted approach to identify specific small molecules in plasma as candidate biomarkers of insufficient sleep. Investigators will conduct a controlled in-laboratory insufficient sleep protocol where participants receive 2 days of 5 hour sleep opportunities per night on 2 separate occasions. Plasma will be collected for metabolomics analyses every 2 hours (across 24 hours) during scheduled wakefulness at baseline and during insufficient sleep. Participants will complete the insufficient sleep protocol twice, separated by 23 days of sufficient sleep, to identify which plasma metabolites consistently change during insufficient sleep. Investigators anticipate these findings will be the first step in establishing validated biomarkers of impaired sleep that will advance our understanding, assessment and management of health consequences and symptoms associated with insufficient sleep.

ELIGIBILITY:
Inclusion Criteria:

* normal Body mass index (18.5-24.9)
* normal blood chemistries
* habitual sleep duration ~7 - 9.25 hours
* live at Denver altitude or higher for at least 3 months

Exclusion Criteria:

* must not be participating in another research study that could influence safe participation in the current study
* any clinically significant medical or surgical condition within last year
* clinically significant abnormality during physical examination
* any physician determined significant abnormality in vital signs, EKG, or clinical laboratory values
* any clinically significant psychiatric condition defined by DSM-V
* any clinically significant sleep disorder
* use of medications/supplements/drugs within one month of study or need of medications during study
* symptoms of active illness
* uncorrected visual impairment
* working shift-work in year prior to study
* travel more than 1 time zone in 3 weeks prior to study
* pregnant/nursing
* greater than moderate caffeine or alcohol use
* positive toxicology screening
* current smoker

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Plasma Metabolomics Biomarker Fingerprint | Plasma will be collected for metabolomics analyses every 2 hours during scheduled wakefulness at baseline and during the final 24 hours of insufficient sleep for both visits one and two
  Investigators can detect ~4,000 plasma metabolites and will identify which metabolites have consistent, sensitive, and specific responses to insufficient sleep across visits one and two. These metabolites will be identified as candidate biomarkers of insufficient sleep.

SECONDARY OUTCOMES:
Psychomotor Vigilance Test | Participants will complete the psychomotor vigilance test every 3 hours during scheduled wakefulness across baseline and insufficient sleep for visits one and two
  The Psychomotor Vigilance Test is a reaction time based test designed to evaluate the ability to sustain attention.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth P Wright, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- Sleep and Chronobiology Laboratory, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data generated from the proposed work that is presented in a peer reviewed journal will be uploaded, de-identified, into the Metabolomics Data Repository and Coordinating Center (DRCC) (U01) through UCSD; http://www.metabolomicsworkbench.org/nihmetabolomics/datasharing.html. In addition, .raw data that is presented in a peer reviewed journal will be archived indefinitely and made available upon request.